CLINICAL TRIAL: NCT01907230
Title: Propylactic Use of Entecavir for Biological Agents Associated Hepatitis B Virus Reactivation in Inflammatory Arthritis Patients: a Randomized Controlled Trial
Brief Title: Entecavir for Biological Agents Associated HBV Reactivation in Inflammatory Arthritis Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Professor: Yi-Hsiang Huang, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AI463-962
Record Dates: First submitted 2013-07-14; First posted 2013-07-24 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Rheumatoid Arthritis; Hepatitis B Reactivation; Exposure to Hepatitis B Virus
Keywords: Rheumatoid arthritis; Inactive HBV carrier; Resolved Hepatitis B; HBV reactivation; Anti-tumor necrotic factor-alfa
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Entecavir, Prophylactic group (Experimental): Participants will initiate entecavir 0.5 mg/day orally one week before biologic treatment. Entecavir treatment will be continued normally for 12 months (6 months after stopping biologic therapy or till restart another course of biologic treatment if the clinicians' judgment is minimal risk of reactivation after the first course of biologic agent treatment).
  Interventions: Drug: Entecavir
- Control group (pre-emptive treatment) (No Intervention): Patients will start entecavir therapy, 0.5 mg/day orally, when reactivation of HBV (defined as detectable HBV viral loads for 2 consecutive visits with at least one month apart), and continued entecavir treatment until undetectable HBV viral loads for 1 year (consistent with current APASL recommendation).

INTERVENTIONS:
Drug: Entecavir — In the prophylactic group, participants will initiate entecavir 0.5 mg/day orally one week before biologic treatment. Entecavir treatment (adjust dosage according to renal function) will be continued normally for 12 months (6 months after stopping biologic therapy or till restart another course of biologic treatment if the clinicians' judgment is minimal risk of reactivation after the first course of biologic agent treatment).
  Other Names: Baraclude
  Arms: Entecavir, Prophylactic group

SUMMARY:
Antiviral prophylaxis can prevent the risk of biologic agents-associated HBV reactivation in hepatitis B inactive carriers and patients with past HBV infection

DETAILED DESCRIPTION:
The risk of HBV reactivation is associated with the intensity of immunosuppression. Biological therapies block the action of biological products involved in immune-inflammatory pathogenesis of many diseases. However, these biologic agents induce a profound immunosuppression, and their use has been reported to be associated with HBV reactivation. Currently, the actual incidence of HBV reactivation in inflammatory arthritis patients who underwent biologic treatments (TNF-α blockades) is unclear, especially in inflammatory arthritis (IA) patients with past hepatitis B infection. In this study, we plan to enroll IA patients who are inactive HBV carriers (HBsAg-positive/ HBV viral loads <2000 IU/ml; subgroup 1), or have past HBV infection (HBsAg-negative/anti-HBc-positive/ HBV viral loads < 2000 IU/ml; subgroup 2); and first line biologic treatment (Humira or Enbrel or Simponi or Orencia or Mabthera or Actemra) is indicated. Patients will be randomized in a 1:1 ratio to receive either prophylactic or therapeutic entecavir treatment for each subgroup. In the prophylactic group, participants will initiate entecavir 0.5 mg/day orally one week before biologic treatment. Entecavir treatment will be continued normally for 12 months. In the therapeutic group, patients will start entecavir therapy, 0.5 mg/day orally, when reactivation of HBV (pre-emptive treatment). HBV reactivation is defined as HBV viral loads > 2,000 IU/ml for 2 consecutive visits of one month apart. The main goal of the study is to delineate the incidence of HBV reactivation during and after biologic treatment in IA patients who are inactive HBV carriers or have past HBV infection, and tries to define the optimal HBV monitoring and antiviral prophylactic strategy in IA patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age : from 20 to 90 y/o.
2. HBsAg-positive for more than 6 months and HBV DNA < 2000 IU/ml (Subgroup 1）or HBsAg-negative but anti-HBc positive with HBV DNA < 2000 IU/ml (Subgroup 2）.
3. Inflammatory arthritis patients who plan to treat with biological agents, including Humira or Enbrel or Simponi or Orencia or Mabthera or Actemra; as first line biologic treatment is indicated.

Exclusion Criteria:

1. HCV, HIV, or HDV coinfection.
2. Uncontrolled HCC or other malignancy within 3 years.
3. Decompensated liver cirrhosis (CTP score ≥ 7).
4. Uremia patients under hemodialysis or continuous ambulatory peritoneal dialysis or patients with Ccr < 50 mL/min
5. Pregnant or breastfeeding women.
6. Women of child-bearing potential (WOCBP) who are unwilling or unable to use an acceptable method of contraception to avoid pregnancy throughout the study and for up to 4 weeks after the last dose of study drug.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2013-09-10 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
HBV reactivation | 12 months after biologic treatment
  The main goal of the study is to delineate the incidence of HBV reactivation during and after biologic treatment in IA patients who are inactive HBV carriers or have past HBV infection, and tries to define the optimal HBV monitoring and antiviral prophylactic strategy in IA patients.

SECONDARY OUTCOMES:
HBsAg reverse seroconversion in occult HB patients. | 12 months after biologic treatment
Hepatitis flare (ALT > 100 U/L) related to biological treatments | 12 months after biologic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Hsiang Huang, MD, Ph.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Division of Gastroenterology & Division of Allergy Immunology and Rheumatology, Taipei Veterans General Hospital, Taipei, Taiwan